CLINICAL TRIAL: NCT06568614
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of BG-89894 (SYH2039) Tablets in Patients With Advanced Solid Tumors
Brief Title: An Investigational Study of BG-89894 Tablets in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG-89894-101; SYH2039-001 (Other: BeOne); CTR20242626 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Advanced or Metastatic MTAP-deleted Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a: Dose Escalation and Safety Expansion (Experimental): Sequential cohorts of increasing dose levels of BG-89894 (SYH2039) will be evaluated as monotherapy.
  Interventions: Drug: BG-89894
- Phase 1b: Dose Expansion and Optimization (Experimental): Multiple indication-specific cohorts will be evaluated for safety, tolerability, and potential dose optimization of BG-89894 (SYH2039).
  Interventions: Drug: BG-89894

INTERVENTIONS:
Drug: BG-89894 — Administered orally
  Other Names: SYH2039

SUMMARY:
This study is being done to learn more about a new drug called BG-89894 (previously known as SYH2039). Researchers want to see if the drug is safe, how well people can tolerate it, how it moves through the body, and whether it shows any early signs of helping to treat cancer. The information gathered may help guide how future studies are designed. The entire study is expected to last about four years. People who join the study may receive treatment for around six months and will be followed for about 12 months after their treatment ends. The study plans to enroll participants over a three-year period.

ELIGIBILITY:
Key Inclusion Criteria:

* Must sign a written informed consent and willing to comply with all study-related procedures and requirements.
* Age ≥18 years (or the legal age of consent according to local regulations).
* Histologically or cytologically confirmed diagnosis of advanced, metastatic, or unresectable solid tumors that have progressed on or after standard therapy, or for which no appropriate standard therapy is available.
* Evidence of Methylthioadenosine phosphorylase (MTAP) homozygous deletion or loss of MTAP expression in tumor tissue.
* Participants must be able to provide an archived tumor tissue sample or unstained fresh biopsy if there is no archival tissue at baseline.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and evidence of adequate organ function and bone marrow reserve, as defined in the study protocol.

Key Exclusion Criteria:

* History of other malignancies or concurrent active malignancies within 3 years.
* Prior treatment with methionine adenosyltransferase 2 alpha (MAT2A) inhibitors (e.g., AG-270, IDE397) or methylthioadenosine (MTA)-cooperative protein arginine methyltransferase 5 (PRMT5) inhibitors (e.g., AMG193).
* Uncontrolled or active central nervous system (CNS) disease, including untreated or symptomatic brain metastases, spinal cord compression, or leptomeningeal carcinomatosis.
* Active bleeding, history of major bleeding events within the past 6 months, or tumors associated with a high risk of vascular invasion.
* Receipt of systemic anticancer therapy, radiation therapy, live vaccine, or major surgical procedures within protocol-specified washout periods.
* Active or uncontrolled infections, including tuberculosis (TB), (COVID-19, known human immunodeficiency virus (HIV) infection, or uncontrolled hepatitis B virus (HBV) infection.

Note: Additional eligibility criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-10-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From first dose of the study drug to 30 days after the last dose or initiation of a new anticancer therapy, whichever occurs first (approximately 18 months)
  Number of participants experiencing adverse events and serious adverse events as determined per Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0), including findings from physical examinations, electrocardiograms (ECGs), laboratory assessments, and that meet protocol-defined dose-limiting toxicity (DLT) criteria.
Phase 1a: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) | Approximately 1 month
  MTD is defined as the highest dose evaluated for which estimated toxicity rate is the closest to the target toxicity rate. MAD is defined as the highest dose administered if MTD is not reached.
Phase 1a: Recommended dose(s) for expansion (RDFE) of BG-89894 | Approximately 18 months
  RDFE is defined as dose level(s) recommended for expansion that will be determined based on the MTD or MAD, taking into consideration the longterm tolerability, pharmacokinetics, pharmacodynamics, preliminary antitumor activity, and any other relevant data, as available.
Phase 1b: Recommended Phase 2 Dose (RP2D) | Approximately 18 months
  R2PD is defined as the dose level recommended for phase 2 that will be determined based on safety, tolerability, pharmacokinetics, pharmacodynamics, preliminary antitumor activity, and other relevant data.
Phase 1b: Overall Response Rate (ORR) | Approximately 18 months
  ORR is defined as the percentage of participants who had confirmed complete response (CR) or partial response (PR) as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Phase 1a and 1b: Maximum observed plasma concentration (Cmax) of BG-89894 | Twice in the first month
Phase 1a and 1b: Time to reach maximum observed plasma concentration (Tmax) of BG-89894 | Twice in the first month
Phase 1a and 1b: Apparent terminal elimination half-life (t1/2) of BG-89894 | Twice in the first month
Phase 1a and 1b: Apparent volume of distribution (Vd/F) of BG-89894 | Twice in the first month
Phase 1a and 1b: Apparent total clearance (CL/F) of BG-89894 | Twice in the first month
Phase 1a and 1b: Area under the concentration-time curve (AUC) for BG-89894 | Twice in the first month
Phase 1b: Minimum observed plasma concentration (Cmin) of BG-89894 | Approximately up to 6 months
Phase 1b: Accumulation Ratio (AR) of BG-89894 | Twice in the first month
Phase 1a: Overall response rate (ORR) | Approximately 18 months
  ORR is defined as the percentage of participants who had confirmed complete response (CR) or partial response (PR) as assessed by the investigator per RECIST v1.1.
Phase 1a and 1b: Duration of response (DOR) | Approximately 18 months
  DOR is defined as the time from the first determination of objective response that is confirmed until the first documentation of disease progression or death, whichever comes first as assessed according to RECIST v1.1 by the investigator.
Phase 1a and 1b: Disease Control Rate (DCR) | Approximately 18 months
  DCR is defined as the percentage of participants with the best overall response of confirmed CR, PR, or stable disease as assessed according to RECIST v1.1 by the investigator.
Phase 1b: Progression free survival (PFS) | Approximately 18 months
  PFS is defined as the time from the date of the first dose of study drug to the date of the first documentation of disease progression assessed by the investigator using RECIST v1.1 or death, whichever occurs first.
Phase 1b: Number of particpants with AEs and SAEs | From first dose of the study drug to 30 days after the last dose or initiation of a new anticancer therapy, whichever occurs first (approximately 24 months)
  Number of participants experiencing adverse events and serious adverse events as determined per CTCAE v5.0, including findings from physical examinations, ECGs, and laboratory assessments as needed.
Phase 1b: Plasma Concentrations | Approximately up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (20):
- United States (4):
  - Sidney Kimmel Comprehensive Cancer At Johns Hopkins, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - Next Virginia, Fairfax, Virginia
- Australia (4):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Cancer Research South Australia, Adelaide, South Australia
  - St Vincents Hospital, Fitzroy, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- China (12):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial Peoples Hospital Huifu Branch, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Hospital of China Medical University Hunnan Branch, Shenyang, Liaoning
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials